CLINICAL TRIAL: NCT00729638
Title: An Open-Label Phase I Study of the Safety of and Efficacy of RAD001 in Combination With Lenalidomide in the Treatment of Subjects With Relapsed and Relapsed/Refractory Multiple Myeloma
Brief Title: RAD001 and Lenalidomide in the Treatment of Subjects With Relapsed and Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Mayo Clinic (Other); Memorial Sloan Kettering Cancer Center (Other); Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Noopur Raje, Director, Center for Multiple Myeloma, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-288; RV-MM-PI-142
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Multiple Myeloma
Keywords: relapsed multiple myeloma; refractory multiple myeloma; RAD001; lenalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — Everolimus; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): Single arm phase I study
  Interventions: Drug: RAD001; Drug: lenalidomide

INTERVENTIONS:
Drug: RAD001 — Dose levels will change: Taken orally either every other day for the first three weeks of each cycle or taken every day for the first three weeks of each cycle.
Drug: lenalidomide — Dose level will vary: taken orally 30-60 minutes after taking RAD001 every day for the first three weeks of each cycle.

SUMMARY:
The purpose of this research study is to determine the highest dose of lenalidomide and RAD001 that can be given without causing too many serious side effects. Another goal of this research study is to look at how the participants cancer may respond to the study treatment. Additionally, we wish to learn more about how the body breaks down and gets rid of the study drugs. We will also try to find substances in the blood (biomarkers) that may help predict how myeloma will respond to study treatment.

DETAILED DESCRIPTION:
* Researchers are looking for the highest doses of RAD001 and lenalidomide used in combination that can be given safely so small groups of people will be enrolled in steps in this trial. The first group will be given a certain dose of RAD001 and a certain dose of lenalidomide. If they have few or manageable side effects, the next small group of people will be enrolled with a higher dose of RAD001 and/or a higher dose of lenalidomide. This will continue until the highest dose of the drugs used is determined.
* Study treatment will be given in 28 day cycles. Both RAD001 and lenalidomide are pills that are taken orally. Both drugs will be started on the same day. RAD001 will be taken either every other day or every day for the first 3 weeks (days 1-21) of each 28-day cycle. Lenalidomide will be taken daily for the first 3 weeks (days 1-21) of each cycle.
* Participants will come to the clinic weekly during the first cycle to monitor side effects. The following will be performed at these clinic visits: physical examination, medical history update, questionnaires, and blood work.
* On cycles 2-8, participants will come to the clinic on Day 1 of each cycle. The following will be performed at this clinic visit: physical examination, medical history update, questionnaire, and blood word.
* At the end of cycle 8, a skeletal survey, bone marrow aspiration and biopsy will be performed to check response to study treatment.
* Participants may continue to receive RAD001 and lenalidomide beyond 8 cycles if their cancer does not get worse and they do not have unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Subject was previously diagnosed with multiple myeloma bases on standard criteria listed in protocol
* Patients must have relapsed or relapsed/refractory disease
* 18 years of age or older
* All necessary baseline studies for determining eligibility must be obtained within 21 days prior to enrollment
* ECOG Performance Status of 0 to 2
* Able to take aspirin (81 or 325mg) daily as prophylactic anticoagulation
* Prior thalidomide/lenalidomide therapy is allowed
* Able to take bactrim
* Female of childbearing potential must have a negative serum or urine pregnancy test

Exclusion Criteria:

* Renal insufficiency
* Concommitant therapy medications that include corticosteroids or other chemotherapy that is or may be active against myeloma or therapy with chemotherapy within 2 weeks prior to day 1. Nitrosoureas must be discontinued 6 weeks prior to day 1. Concurrent radiation therapy is not permitted.
* Subjects with evidence of mucosal or internal bleeding and/or platelet refractory
* Subjects with poorly controlled diabetes mellitus
* Subjects with an ANC < 10-00 cells/mm3
* Subjects with a hemoglobin < 8.0 g/Dl
* AST (SGOT and ALT (SGPT) greater or equal to 2x ULN
* Prior therapy with RAD001
* Known hypersensitivity to thalidomide or lenalidomide
* Any condition, including laboratory abnormalities, that in the opinion of the Investigator, places the subject at unacceptable risk if he/she were to participate in the study
* Clinically relevant active infection or serious co-morbid medical conditions such as recent thromboembolic disease are ineligible if occurred less than 2 weeks prior to enrollment or clinically unstable
* Chronic obstructive or chronic restrictive pulmonary disease, difficult to control diabetes, upper gastrointestinal ulceration, and cirrhosis
* Prior malignancy (within the last 3 years) except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, in situ prostate cancer or other cancer for which the subject has been disease-free for at least 3 years
* Pregnant or breast-feeding females
* Prior treatment with any investigational drug within preceding 4 weeks
* Major surgery, and or radiation with 2 weeks of study initiation
* Uncontrolled leptomeningeal disease
* Prior treatment with other mTOR inhibitors
* The use of G-CSF is not permitted to render the patient eligible fot the study
* POEMS syndrome
* Known HIV infection
* Known active Hepatitis B or C infection
* Myocardial infarction within 6 months prior to enrollment or has NYHA Class III or IV heart failure, uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001
* Patients with active, bleeding diathesis or on oral anti-vitamin K medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of RAD001 when given in combination with lenalidomide and to identify the maximum tolerated dose (MTD) as well as a recommended Phase 2 dose for the combination in this patient population. | 2 years

SECONDARY OUTCOMES:
To evaluate the response to the combination of RAD001 and lenalidomide in subjects with multiple myeloma. | 2 years
To determine the pharmacokinetics of RAD001 and lenalidomide. | 2 years
To identify possible surrogate markers to better define mechanisms of action for the combination of the two drugs. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Noopur Raje, MD, Principal Investigator — Massachusetts General Hospital
Locations (5):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Result] Yee AJ, Hari P, Marcheselli R, Mahindra AK, Cirstea DD, Scullen TA, Burke JN, Rodig SJ, Hideshima T, Laubach JP, Ghobrial IM, Schlossman RL, Munshi NC, Anderson KC, Weller EA, Richardson PG, Raje NS. Outcomes in patients with relapsed or refractory multiple myeloma in a phase I study of everolimus in combination with lenalidomide. Br J Haematol. 2014 Aug;166(3):401-9. doi: 10.1111/bjh.12909. Epub 2014 Apr 25. PMID 24761838